CLINICAL TRIAL: NCT01314469
Title: Influence of Macular Edema on Quality of Life in Patients With Non-infectious Intermediate Uveitis
Brief Title: Quality of Life in Patients With Intermediate Uveitis
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Other Study IDs: 2008-559-f-S
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-03

CONDITIONS: Macular Edema
Keywords: Quality of life in patients with macular edema compared to patients without macular edema.
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients with intermediate uveitis

SUMMARY:
The aim of this study is to determine if macular edema is associated with less visual function and quality of live in patients with intermediate uveitis

ELIGIBILITY:
Inclusion Criteria:

* Pars planitis

Exclusion Criteria:

* Patients with any other diseases
* Patients under age 18

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate uveitis
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology at St Franziskus Hospital, Münster, Germany